CLINICAL TRIAL: NCT06999603
Title: A Phase 2, Two-part Study to Assess the Safety, Antiviral Biomarker Responses, and Efficacy of Inhaled SNG001 for the Treatment of Patients With a Confirmed Respiratory Virus Infection Undergoing Invasive Mechanical Ventilation
Brief Title: Phase 2 Study of Inhaled SNG001 in Mechanically Ventilated Patients With Respiratory Viral Infection
Acronym: INVENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Synairgen Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SG021; 2024-520375-27-00 (EU CTIS Number); U1111-1317-0525 (Other: WHO); ISRCTN30482473 (Other: ISRCTN)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Viral Pneumonia
Keywords: Influenza; Respiratory Syncytial Virus; Rhinovirus; Adenovirus; Human Metapneumovirus; Coronavirus; Intubated; Mechanically ventilated; Interferon; Intensive care; SARS-CoV-2; Parainfluenza
MeSH Terms: conditions — Pneumonia, Viral; Influenza, Human; Adenoviridae Infections; Coronavirus Infections; Paramyxoviridae Infections

STUDY DESIGN:
Intervention Model Description: Part 1 of this study will include a low-dose (one syringe) first cohort, followed by an optional second cohort utilising a two-syringe dose. Part 2 will commence following the conclusion of Part 1 and will utilise the two-syringe dose. Both Part 1 and Part 2 of the study will be randomised, double-blind and placebo-controlled.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Safety Evaluation of SNG001 (Experimental): Participants will inhale a dose of SNG001 via the Solo nebuliser, once a day for up to 14 days. A first, single syringe, low-dose cohort may be followed by an optional second cohort utilising a two-syringe dose.
  Interventions: Drug: SNG001
- Part 1 Safety Evaluation of SNG001 (Placebo) (Placebo Comparator): Participants will inhale a dose of placebo matched to SNG001 (only excipients of the SNG001 solution) via the Solo nebuliser, once a day for up to 14 days.
  Interventions: Drug: Placebo
- Part 2 Efficacy Evaluation of SNG001 (Experimental): Participants will inhale the higher (two-syringe) dose of SNG001 via the Solo nebuliser, once a day for up to 14 days.
  Interventions: Drug: SNG001
- Part 2 Efficacy evaluation of SNG001 (Placebo) (Placebo Comparator): Participants will inhale a dose of placebo matched to SNG001 (only excipients of the SNG001 solution) via the Solo nebuliser, once a day for up to 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNG001 — SNG001 nebuliser solution is presented as a ready-to-use aqueous solution (neutral pH) in glass syringes containing 0.65 mL of drug product solution containing 12 MIU/mL of IFNβ 1a.
  Arms: Part 1 Safety Evaluation of SNG001; Part 2 Efficacy Evaluation of SNG001
Drug: Placebo — The placebo nebuliser solution is presented in glass syringes containing 0.65 mL of solution containing the same formulation as the study medication but without IFNβ 1a (i.e., only the excipients of the SNG001 solution).
  Arms: Part 1 Safety Evaluation of SNG001 (Placebo); Part 2 Efficacy evaluation of SNG001 (Placebo)

SUMMARY:
The goal of this Phase 2 study is to assess about the safety, antiviral biomarker responses and efficacy of SNG001 when given to patients requiring invasive mechanical ventilation due to a respiratory virus infection. Its ability to speed up virus clearance and reduce mortality, compared with standard of care, will be studied.

The study is split into two parts. All participants will receive standard of care in addition to SNG001 or placebo.

In Part 1, the safety of SNG001 will be assessed. Participants of 50 years and older will receive study drug or placebo once a day for up to 14 days, whilst in hospital.

In Part 2, the primary objective will be the efficacy of SNG001. Participants between 18 and 50 years with an immunocompromising condition and patients over 50 years (with or without an immunocompromising condition) will receive study drug once a day for up to 14 days, whilst in hospital.

ELIGIBILITY:
Part 1 Inclusion Criteria:

To be eligible for randomisation into Part 1 of this study, each participant must fulfil the following criteria:

1. Informed consent or legal representative's consent obtained.
2. Patients ≥50 years of age at the time of consent.
3. Patient admitted to the ICU and requiring invasive mechanical ventilation (IMV) due to a respiratory virus infection.
4. Presence of Influenza A (Flu A), Influenza B (Flu B), respiratory syncytial virus (RSV), rhinovirus (RV), adenovirus, parainfluenza, human metapneumovirus (HMPV), or coronaviruses (including SARS-COV-2 and seasonal coronaviruses) in a nose swab sample, confirmed by a positive virus test using a Sponsor approved rapid POC test (e.g., reverse transcription polymerase chain reaction [RT-PCR]).
5. Time from intubation to administration of first dose of study medication ≤48 hours.
6. Women of childbearing potential must have a negative pregnancy test. For this study, women of childbearing potential are defined as women <55 years old.

Part 1 Exclusion Criteria:

A participant must not be randomised into Part 1 of the study if they meet any of the following criteria:

1. Expected termination of IMV within 24 hours from the time of randomisation
2. Life expectancy <24 hours.
3. Liver failure (Child-Pugh C).
4. Severe congestive heart failure (New York Heart Association [NYHA] IV).
5. Receipt of lung transplant.
6. Known or suspected active tuberculosis, or infection with other mycobacteria
7. Known or suspected active systemic fungal infection.
8. Anticipated transfer to another hospital which would prevent the participant from continuing in the study and completing protocol assessments.
9. Need for long-term mechanical ventilation prior to ICU admission.
10. Use of inhaled sedation.
11. Presence of tracheostomy or laryngectomy.
12. Requirement for airway pressure release ventilation mode.
13. History of hypersensitivity to natural or recombinant IFNβ or to any of the excipients in the drug preparation.
14. Any condition, including findings in the patient's medical history or in the pre-randomisation study assessments that in the opinion of the Investigator, constitute a risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation.
15. Participation in previous clinical studies of SNG001.
16. Current or previous participation in another clinical study where the participant has received a dose of an Investigational Medicinal Product (IMP) containing small molecules within 30 days or 5 half-lives (whichever is longer) prior to entry into this study or containing biologicals within 3 months prior to entry into this study.
17. Known or suspected pregnancy.
18. Females who are breast-feeding or lactating.
19. Immunocompromising condition, including:

    * Established acquired immune deficiency syndrome (AIDS) defined as a cluster of differentiation 4 (CD4) count <200 cells/microL, and/or the presence of any AIDS-defining condition;
    * Haematological malignancy;
    * Bone marrow transplantation; or
    * Immunosuppressive therapy, including:
    * Cancer therapy (e.g. chemo-, radio-, immuno-, hormone or other types of therapy), immune-cell depleting therapy, immunosuppressive therapy for autoimmune disorders, medications for prevention of organ transplantation rejection, administered within 6 months prior to randomisation; or
    * Corticosteroids >20 mg of prednisone or equivalent per day administered continuously for >14 days prior to randomisation.
20. Severe chronic lung disease requiring home oxygen therapy, including chronic obstructive pulmonary disease, asthma, cystic fibrosis, or pulmonary fibrosis.

Part 2 Inclusion Criteria:

To be eligible for randomisation into Part 2 of this study, each participant must fulfil the following criteria:

1.a Patients ≥18 and <50 years of age at the time of consent, with an immunocompromising condition, including:

* Solid tumour malignancy undergoing cancer therapy (e.g. chemo-, radio-, immuno-, hormone or other types of therapy);
* Haematological malignancy in remission, with or without maintenance therapy;
* Immunosuppressive therapy for autoimmune disease;
* Therapy for prevention of organ transplant rejection;
* Corticosteroids >20 mg of prednisone or equivalent per day, administered continuously for >14 days prior to randomisation or

  1. b Patients ≥50 years of age at the time of consent, with or without an immunocompromising condition (as defined above).
  2. Patient admitted to the ICU and requiring IMV due to a respiratory virus infection.
  3. Presence of Flu A, Flu B, RSV, RV, adenovirus, parainfluenza, HMPV, or coronaviruses (including SARS-COV-2 and seasonal coronaviruses) in a Lower Respiratory Tract sample, confirmed by a positive virus test using a Sponsor approved rapid POC test (e.g., RT-PCR).
  4. Time from intubation to administration of first dose of study medication ≤48 hours.
  5. Informed consent or legal representative's consent obtained.
  6. Women of childbearing potential must have a negative pregnancy test. For this study, women of childbearing potential are defined as women <55 years old.

Part 2 Exclusion Criteria:

A participant must not be randomised into Part 2 of the study if they meet any of the following criteria:

1. Expected termination of IMV within 24 hours from the time of randomisation.
2. Life expectancy <24 hours.
3. Liver failure (Child-Pugh C).
4. Severe congestive heart failure (NYHA IV).
5. Receipt of lung transplant.
6. Known or suspected active tuberculosis, or infection with other mycobacteria.
7. Known or suspected systemic fungal infection.
8. Immunocompromising condition, including:

   * Haematological malignancy requiring induction or consolidation therapy within 3 months prior to randomisation;
   * Bone marrow transplant within 6 months prior to randomisation;
   * Solid organ transplant within 6 months prior to randomisation;
   * Corticosteroids >75 mg of prednisone or equivalent per day, administered continuously for >7 days prior to randomisation;
   * Methotrexate therapy at randomisation, if the indication is chemotherapy for cancer;
   * Chimeric antigen receptor (CAR)-T cell therapy, administered within 3 months prior to randomisation;
   * Ibrutinib or alemtuzumab, administered within 3 months prior to randomisation;
   * Neutropenia <500/mm3 not due to sepsis;
   * Clinical presentation consistent with severe bone marrow suppression or pancytopenia;pancytopenia;
   * Established AIDS, defined as a CD4 count <200 cells/microL, and/or the presence of any AIDS-defining condition.
9. Anticipated transfer to another hospital which would prevent the participant from continuing in the study and completing protocol assessments.
10. Need for long-term mechanical ventilation prior to ICU admission.
11. Use of inhaled sedation.
12. Presence of tracheostomy or laryngectomy
13. History of hypersensitivity to natural or recombinant IFNβ or to any of the excipients in the drug preparation.
14. Any condition, including findings in the patient's medical history or in the pre-randomisation study assessments that in the opinion of the Investigator, constitute a risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation.
15. Participation in previous clinical studies of SNG001.
16. Current or previous participation in another clinical study where the participant has received a dose of an IMP containing small molecules within 30 days or 5 half-lives (whichever is longer) prior to entry into this study or containing biologicals within 3 months prior to entry into this study.
17. Known or suspected pregnancy.
18. Females who are breast-feeding or lactating.
19. Severe chronic lung disease requiring home oxygen therapy, including chronic obstructive pulmonary disease, asthma, cystic fibrosis, or pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Part 1: AE and SAE Severity | Up to 28 days from randomisation
  The occurrence and severity of AEs and serious adverse events (SAEs), including pre-specified respiratory and cardiovascular deteriorations.
Part 2: All-cause mortality | Within 28 days from randomisation
  All deaths recorded on study

SECONDARY OUTCOMES:
Part 2: AE and SAE severity | Up to 42 days from randomisation
  The occurrence and severity of AEs and SAEs, including pre-specified respiratory and cardiovascular deteriorations.
Part 2: Change in mSOFA from baseline | Up to 14 days
  Change from baseline in modified Sequential Organ Failure Assessment (mSOFA) score during ICU (intensive Care Unit) stay.
Part 2: Time to Extubation | Up to 28 days from randomisation
  Time to extubation.
Part 2: Number of ventilator free days | Up to 28 days from randomisation
  Ventilator-free days over 28 days from randomisation
Part 2: Duration of stay in ICU | Up to 28 days from randomisation
  Duration of ICU stay.
Part 2: Duration of stay in hospital | Up to 28 days from randomisation
  Duration of hospital stay.
Part 2: Change in OSCI from baseline | Up to 28 days from randomisation
  Change in Ordinal Scale for Clinical Improvement (OSCI) score from baseline to 7, 10, 14 and 28 days post randomisation.
Part 2: Time to first negative virus test | Up to 14 days from randomisation
  Time to first negative virus test in tracheal aspirates.
Part 2: Change in IFNβ levels from baseline | Up to 14 days from randomisation
  Change from baseline in levels of IFNβ dependent biomarkers in tracheal aspirates
Part 2: No organ support | At 28 days from randomisation and at 28 days post final dose
  Alive and free of organ support
Part 2: All Cause Mortality | Within 28 days post final dose
  All deaths recorded post final dose

CONTACTS AND LOCATIONS:
Locations (67):
- United States (22):
  - University of California - Davis, Sacramento, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - NCH Pulmonary Critical Care, Naples, Florida
  - Emory University, Atlanta, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Sinai-Grace Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - VA Western New York Healthcare system, Buffalo, New York
  - NYU Langone Tisch Hospital, New York, New York
  - University of North Carolina (UNC), Chapel Hill, North Carolina
  - University of Cincinnati Medical Center (UCMC), Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University (OSU), Columbus, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - AnMed Health Pulmonary and Sleep Medicine, Anderson, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (4):
  - Universitair Ziekenhuis Brussel, Brussels
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - Centre Hospitalier Régional de la Citadelle, Liège
  - Centre Hospitalier Universitaire (CHU) de Liege, Liège
- France (12):
  - Centre Hospitalier d'Argenteuil, Argenteuil
  - Centre Hospitalier de Bourg-en-Bresse, Bourg-en-Bresse
  - CHD Vendee, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CHU de Lille, Lille
  - CHU de Limoges - Hopital Dupuytren 1, Limoges
  - CHU de Nantes - Hotel-Dieu, Nantes
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rouen - Hopital Charles-Nicolle, Rouen
  - CHU St Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - CHRU de Strasbourg, Strasbourg
  - CHRU de Tours - Hopital Bretonneau, Tours
- Netherlands (4):
  - Ziekenhuis Gelderse Vallei, Ede
  - Canisius-Wilhelmina Ziekenhuis (CWZ), Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari Mutua Terrassa, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (20):
  - Torbay Hospital, Paignton, Devon
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Royal Sussex County Hospital, Brighton
  - Cardiff and Vale Hospital, Cardiff
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - Leicester Royal Infirmary, Leicester
  - University College London Hospital, London
  - Royal Free Hospital, London
  - St George's Hospital, London
  - Manchester Royal Infirmary, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Queens Medical Centre (QMC), Nottingham
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided